CLINICAL TRIAL: NCT07270536
Title: The Impact of Accelerated Pacing and AV-delay Regulation on the Pulmonary Capillary Wedge Pressure During Exercise in Patients With HFpEF
Brief Title: Accelerated Pacing and Cardiac Filling Pressures During Exercise in Patients With Heart Failure With Preserved Ejection Fraction
Acronym: APAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Jessa Ziekenhuis Hasselt (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S70922
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: HFpEF
Keywords: Heart Failure with Preserved Ejection Fraction; Accelerated pacing; Chronotropic response; Hemodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental)
  Interventions: Other: Accelerated pacing with AV-delay optimization during rest and light intensity cycling

INTERVENTIONS:
Other: Accelerated pacing with AV-delay optimization during rest and light intensity cycling — Patients will undergo one protocol at rest and two exercise protocols (10 Watts followed by 25 Watts). During each protocol, the pacemaker rate will be gradually increased in three stages. At each stage, intracardiac pressures and shear-wave velocity will be measured. In a final fourth stage, the pacemaker rate will return to the level associated with the lowest heart pressure, blood oxygen levels and oxygen uptake will be assessed.

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a condition where the heart pumps strongly enough, but has trouble relaxing and filling with blood properly. This causes the pressure on the left side of the heart to rise, especially during activity, which can lead to symptoms like shortness of breath and fatigue. Even light activities such as walking or climbing stairs can be difficult, limiting daily life.

Recent research suggests that increasing the heart rate in people with HFpEF may help lower this elevated pressure in the heart. Because patients usually experience their symptoms during exercise, this study aims to see whether, during light activity, increasing the heart rate in patients who already have a pacemaker by adjusting its settings, can reduce this elevated pressure in the heart. Furthermore, we will look at how increasing the heart rate affects the amount of blood the heart pumps each minute, another key factor in a person's ability to perform physical activity.

The investigators will examine 20 patients using a heart catheter to measure pressures, along with breathing analyses. During the measurements, all patients will perform light-intensity cycling.

If increasing the pacemaker rate lowers the pressure in the heart, this simple, non-drug-based intervention could improve daily functioning and comfort for thousands of patients with heart failure, justifying further long-term studies to evaluate effects beyond the immediate changes in heart pressures.

DETAILED DESCRIPTION:
The first phase of the study is the screening phase. During this phase, the investigators will review all patients from the LBBA pacing registries at UZ Leuven and Jessa Hospital to identify who may be eligible. From this review, the investigators will create a list of potential candidates, who will then be contacted during their regular check-up visits, which take place at least once a year. If a patient is found to be eligible during this visit, the study visit will be scheduled within three weeks.

If the patient remains eligible, the study tests will begin. A small tube (catheter) will be placed in a vein in the neck and in an artery in the wrist to measure heart pressures and blood oxygen levels. The patient will then be positioned on a slightly reclined stationary bike. During the test, the heart rate will be gradually increased in three steps by adapting the pacemaker settings, and at each step, the pressures inside the heart will be measured. In a final step, the heart rate will return to the level associated with the lowest heart pressure, and blood oxygen levels will be checked. This allows the research team to calculate how much oxygen the heart pumps per minute.

After the exercise, the patient will rest briefly while the catheters are safely removed.

The entire study visit lasts about three hours, after which participation ends. The full study is expected to be completed once 20 patients have finished all study tests, which should take approximately one year.

ELIGIBILITY:
Participants eligible for inclusion in this study must meet all of the following criteria:

1. Voluntary written informed consent of the participant has been obtained prior to any screening procedures
2. At least 18 years of age at the time of signing the Informed Consent Form (ICF)
3. Heart failure with preserved ejection fraction, defined as one of the below criteria:

   1. HFA-PEFF score >= 5 or
   2. H2FPEF score >= 6 or
   3. EF >= 50% and

   i. Heart failure hospitalization after pacemaker implantation or ii. On loop-diuretics at time of inclusion
4. Having a DDD-pacemaker with LBB area pacing, implanted at least 12 weeks before iCPET
5. >=6 weeks on optimal HFpEF therapy (MRA and SGLT2i), unless contraindicated or not tolerated
6. Sinus rhythm at time of screening and iCPET

Participants eligible for this Study must not meet any of the following criteria:

1. Participant has a history of:

   1. Evidence of significant pulmonary comorbidity based on abnormal pulmonary function tests (FEV1 <60%) or aberrant lung parenchyma more than mild on radiological imaging
   2. Severe/symptomatic valvular diseases
   3. Severe pulmonary hypertension (PASP > 55mmHg estimated by Doppler Echo)
   4. Unstable arrhythmias (VT, VF)
   5. Recurrent syncopes after pacemaker implantation
   6. Episode of atrial fibrillation in the last 3 months
   7. Amyloid cardiomyopathy
2. Physical inability to perform exercise
3. More than 1 hospitalization for heart failure in the last year
4. Resting heart rate> 100bpm
5. At time of iCPET or inclusion: decompensated heart failure, unstable coronary syndrome
6. Contraindication to central venous access

   1. Severe coagulopathy (e.g., spontaneous INR > 2, thrombocytopenia < 50,000/µL)
   2. Local infection or skin infection at the insertion site
   3. Thrombosis or anatomical abnormalities of the right jugular vein
   4. Pneumothorax or contralateral lung pathology
   5. Inability to properly position the patient
7. Contraindication to arterial access

   1. Thrombosis or occlusion of the target artery
   2. Raynaud's phenomenon or other vasospastic disorders
   3. Active infection at the intended insertion site
   4. Severe coagulopathy (e.g., spontaneous INR > 2, thrombocytopenia < 50,000/µL)
   5. Insufficient collateral circulation (e.g., inadequate perfusion in an Allen test)
8. Contraindications to CPET

   1. ECG signifying myocardial injury
   2. ECG signifying current or potentially lethal arrhythmias
   3. Systemic hypotension (e.g. systolic blood pressure < 90 mmHg)
   4. Extreme hypertension (e.g. systolic blood pressure > 220 mmHg)
   5. Syncope, presyncope, or lightheadedness
   6. SaO2 < 88%
   7. Severely elevated PCWP (> 40 mmHg) during exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary capillary wedge pressure (PCWP), measured using a Swan-Ganz catheter (pulmonary artery catheter). | Intraprocedural
  The change in pulmonary capillary wedge pressure at each pacing step compared to the pulmonary capillary wedge pressure at the intrinsic heart rate at rest and during exercise (cycling at 10 Watts and 25 Watts).
  The PCWP at the intrinsic heart rate is defined as the average of the PCWP at the intrinsic heart rate heart rate before and after each pacing step.

SECONDARY OUTCOMES:
Cardiac output, measured using the direct Fick principle | Intraprocedural
  The change in cardiac output (CO), measured by the direct Fick principle, at the pacing frequency corresponding to the greatest reduction in PCWP compared to the intrinsic heart rate at rest and during exercise (cycling at 10 Watts and 25 Watts)
Shear wave velocity, measured via echocardiographically obtained myocardial shear waves following mitral valve closure | Intraprocedural
  The change in shear wave velocity (SWV) at each pacing rate compared to the intrinsic heart rate at rest and during exercise (cycling at 10 Watts and 25 Watts) The shear wave velocity at the intrinsic heart rate is defined as the average of the SWV at the intrinsic heart rate heart rate before and after each pacing step
Peripheral oxygen extraction | Intraprocedural
  The change in peripheral oxygen extraction, measured by the oxygen uptake divided by the cardiac output, at the pacing frequency corresponding to the greatest reduction in pulmonary capillary wedge pressure compared to peripheral oxygen extraction at the intrinsic heart rate at rest and during exercise (cycling at 10 Watts and 25 Watts)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Jessa Ziekenhuis Hasselt, Hasselt
  - University Hospitals Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy considerations and participant confidentiality.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT07270536/Prot_SAP_000.pdf